CLINICAL TRIAL: NCT01209663
Title: Intermediate Care - Effect on Mortality Following Emergency Abdominal Surgery
Acronym: InCare
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: 30th November 2012. Please see breif summary.
Sponsor: Copenhagen University Hospital at Herlev (Other)
Collaborators: University of Copenhagen (Other); Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); Herlev Hospital (Other); Sygekassernes Helsefond (Other); Danish Council for Independent Research (Other); AP Moeller Foundation (Other); Lundbeck Foundation (Other); Hilleroed Hospital (Unknown); Zealand University Hospital (Other); Bispebjerg Hospital (Other); Herning Hospital (Other); Aabenraa Hospital (Other); Vejle Hospital (Other)
Responsible Party: Principal Investigator, Morten Vester-Andersen, MD, Senior resident, Copenhagen University Hospital at Herlev
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-3-2010-010
Record Dates: First submitted 2010-09-24; First posted 2010-09-27 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Emergency Abdominal Surgery
Keywords: General Surgery; Emergency treatment; Postoperative care; Intermediate care unit; High dependency unit; Mortality

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ward Care (Active Comparator): Protocol based discharge to the surgery ward. Observation and treatment is conducted by ward nurses and general surgeons (current treatment).
  Interventions: Other: Postoperative Intermediate Care
- Intermediate Care (Experimental): Observation and treatment in an intermediate care bed in a minimum of 48 hours after randomization. Daily rounds will be carried out by both general surgeons and intensive care physicians.
  Interventions: Other: Postoperative Intermediate Care

INTERVENTIONS:
Other: Postoperative Intermediate Care — Comparison of postoperative Intermediate Care versus Ward Care.
  Other Names: High dependency bed; High dependency unit

SUMMARY:
The objective of this trial is to evaluate postoperative intermediate care versus ward care in patients who have undergone emergency abdominal surgery with a perioperative Acute Physiology and Chronic Health Evaluation (APACHE) II score ≥ 10 (high risk patients).

Patients will be enrolled in the trial, if they are ready to be discharged from the recovery unit or intensive/intermediate care unit to the surgical ward within 24 hours after surgery. Discharge criteria will be according to the Danish national recommendation.

The intermediate care bed in the trial is defined by a certain minimum requirements to patient observation and described treatment possibilities which have to be available to the intermediate bed. If the treatment exceeds these treatment possibilities, the patient will be classified as an intensive care patient. The intermediate care bed will be placed at an intensive care unit, recovery unit or a surgical high dependency unit. If there is no available intermediate care bed, the patients will not be randomized, but only registered as "excluded because of no available intermediate care bed".

Hypothesis: Postoperative intermediate care for 48 hours or more will reduce the 30-day mortality in emergency abdominal surgery patients with a high risk of postoperative organ failure.

Interim analysis: An independent Data Monitoring and Safety Committee (DMSC) will conducted the interim analysis based on the analysis of the primary outcome blinded for intervention allocation. The DMSC will use P<0.001 (Haybittle-Peto) on two subsequent interim analyses as the statistical limit to guide its recommendations regarding early termination of the trial for benefit or harm. The first interim analysis will be conducted when the 30 days follow-up data of about 50% (i.e., about 200 patients) of the trial participants have been obtained and/or 75 deaths have been documented during the trial. If P<0,001 in the first interim analysis a second interim analysis will be conducted when the 30 days follow-up data of about 75% (i.e., about 300 patients) of the trial participants have been obtained and/or 25 deaths have been documented during the trial.

Trial terminated on the 30th November 2012. The Data Monitor Committee found a very low overall event rate of the primary outcome at the first interim-analysis as compared to the pre-trial estimated. This precluding any possibility to detect or reject the anticipated relative risk reduction of 34 % as used in the sample size estimation.

DETAILED DESCRIPTION:
Like Denmark, many European countries has only limited access to surgical intermediate care beds (high dependency beds). This may reflect lack of scientific evidence for the effect of intermediate care combined with restricted healthcare resources. Better access to dedicated postoperative intensive/intermediate care facilities has been suggested as a factor which potentially can reduce postoperative complication rate and mortality in high risk surgical patients. The Incare Trial will provide important data on the effect of postoperative intermediate care in emergency abdominal surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Emergency laparotomy patients treated by general surgeons OR
* Emergency laparoscopic surgery patients treated by general surgeons OR
* Re-operative patients who go through emergency laparotomy or laparoscopy.

AND

* APACHE II score ≥ 10 AND
* Patients who are ready to be discharged to the surgical ward after postoperative stay in the recovering unit or an intermediate/intensive care bed

Exclusion Criteria:

* Appendectomy
* Emergency laparoscopic cholecystectomy
* Emergency diagnostic laparoscopy without intervention
* Postoperative stay in the recovery unit or an intermediate/intensive care bed in more then 24 hours before randomization
* Patients who should not be offered postoperative intensive care
* Patients who have been included in the study earlier
* Age < 18 years
* Trauma patients

Because of slower enrolment rate than anticipated the steering committee have decided on the 3rd of May 2012 to include patients with Apache II score of 10 and 11 although the originally inclusion criteria was Apache II score 12 or above. Patients with Apache II score of 10 and 11 have a high 30 day mortality as well and the potential to benefit from intermediate care. The new criteria was initiated on the 23rd of May 2012 after ethical approval was obtained.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2010-10; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
All cause mortality rate | Within 30 days of surgery

SECONDARY OUTCOMES:
long term mortality | Until 30 days after the last patient is enrolled in the trial
rate of critical care unit admission from ward | Within 30 days of surgery
Postoperative hospitalization time | until 30 days after the last patient is enrolled in the trial

CONTACTS AND LOCATIONS:
Overall Officials: Morten Vester-Andersen, MD, Principal Investigator — Department of Anaesthesiology and Intensive Care Medicine, Copenhagen University Hospital Herlev; Ann M Møller, MD, PhD, Study Chair — Department of Anaesthesiology and Intensive Care Medicine, Copenhagen University Hospital Herlev; Jørn Wetterslev, MD, PhD, Study Chair — Copenhagen Trial Unit, Centre for Clinical Intervention Research, Copenhagen University Rigshospitalet; Jacob Rosenberg, MD, Prof, Study Chair — Department of Gastrointestinal Surgery, Copenhagen University Hospital Herlev; Tina Waldau, MD, PhD, Study Chair — Department of Anaesthesiology and Intensive Care Medicine, Copenhagen University Hospital Herlev; Morten H Møller, MD, PhD, Study Chair — Department of Anaesthesiology and Intensive Care Medicine, Copenhagen University Hospital Bispebjerg; Flemming Moesgaard, MD, PhD, Study Chair — Department of Gastrointestinal Surgery, Copenhagen University Hospital Herlev; Lars N Jørgensen, MD, Prof., Study Chair — Department of Gastrointestinal Surgery, Copenhagen University Hospital Bispebjerg
Locations (7):
- Denmark (7):
  - Copenhagen University, Bispebjerg Hospital, Copenhagen, DK
  - Herning Regional Hospital, Herning, DK
  - Aabenraa Hospital, Aabenraa
  - Herlev University Hospital, Copenhagen
  - Copehagen University, Hilleroed Hospital, Hilleroed
  - Copenhagen University, Koege Hospital, Koege
  - Sygehus Lillebaelt, Vejle Hospital, Vejle

REFERENCES:
- [Derived] Vester-Andersen M, Waldau T, Wetterslev J, Moller MH, Rosenberg J, Jorgensen LN, Jakobsen JC, Moller AM; InCare trial group. Randomized multicentre feasibility trial of intermediate care versus standard ward care after emergency abdominal surgery (InCare trial). Br J Surg. 2015 May;102(6):619-29. doi: 10.1002/bjs.9749. Epub 2015 Mar 18. PMID 25789827
- [Derived] Vester-Andersen M, Waldau T, Wetterslev J, Moller MH, Rosenberg J, Jorgensen LN, Gillesberg I, Jakobsen HL, Hansen EG, Poulsen LM, Skovdal J, Sogaard EK, Bestle M, Vilandt J, Rosenberg I, Berthelsen RE, Pedersen J, Madsen MR, Feurstein T, Busse MJ, Andersen JD, Maschmann C, Rasmussen M, Jessen C, Bugge L, Ording H, Moller AM. Effect of intermediate care on mortality following emergency abdominal surgery. The InCare trial: study protocol, rationale and feasibility of a randomised multicentre trial. Trials. 2013 Feb 2;14:37. doi: 10.1186/1745-6215-14-37. PMID 23374977